CLINICAL TRIAL: NCT00772382
Title: A Phase III, Multi-center, Open Label, Flexible Dose, Long Term Safety Study of MCI-196 in Chronic Kidney Disease Stage V Subjects on Dialysis With Hyperphosphatemia
Brief Title: Study of MCI-196 in Chronic Kidney Disease Stage V Subjects on Dialysis With Hyperphosphatemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tanabe Pharma Corporation (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MCI-196-A06
Record Dates: First submitted 2008-10-10; First posted 2008-10-15 (Estimated); Results first posted 2014-05-12 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Chronic Kidney Disease; Dialysis; Hyperphosphatemia
Keywords: Chronic Kidney Disease; Dialysis; Hyperphosphatemia; Phosphate binder
MeSH Terms: conditions — Renal Insufficiency, Chronic; Hyperphosphatemia | interventions — cholebine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- MCI-196 (Experimental)
  Interventions: Drug: MCI-196

INTERVENTIONS:
Drug: MCI-196 — 3g to 15g/day (3 times a day), Tablet, 52 weeks of flexible dose
  Other Names: Colestilan(INN); Colestimide(JAN); CHOLEBINE®; BindRen®

SUMMARY:
The primary objective of this study is to demonstrate the long-term safety and tolerability of MCI-196 in the subjects with stage V chronic kidney disease on dialysis with hyperphosphatemia.

The secondary objective of this study is to assess the long-term efficacy of flexible doses of MCI-196.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, and is >=18 years old
* Stable hemodialysis or peritoneal dialysis
* Subjects have stable phosphate control
* Subjects on stabilized phosphorus diet
* Subjects undergoing regular dialysis treatment
* Females and of child-bearing potential have a negative serum pregnancy test
* Male subjects must agree to use appropriate contraception

Exclusion Criteria:

* Current clinically significant medical comorbidities, which may substantially compromise subject safety, or expose him/her to undue risk, or interfere significantly with study procedures and which, in the opinion of the Investigator, makes the subject unsuitable for inclusion in the study
* serum albumin level < 3.0g/L
* PTH level > 1000pg/mL
* Hemoglobin level < 8mg/dL
* A History of significant gastrointestinal motility problems
* Biliary obstruction or proven liver dysfunction
* A positive test for HIV 1 and 2 antibodies
* A history of substance or alcohol abuse within the last year
* Seizure disorders
* A history of drug or other allergy
* using cholestyramine, colestipol or colesevelam
* Schedule to receive a kidney transplant within the next 6 months
* Participation in a clinical study with any experimental medication in the last 30 days or an experimental biological product within the last 90 days prior to signing of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2008-12; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Professor, Principal Investigator — Information at Mitsubishi Pharma America
Locations (21):
- United States (17):
  - Los Angeles, California
  - Orange, California
  - Tarzana, California
  - Orlando, Florida
  - Pembroke Pines, Florida
  - Atlanta, Georgia
  - Gurnee, Illinois
  - Evansville, Indiana
  - Baton Rouge, Louisiana
  - New Orleans, Louisiana
  - Northport, New York
  - Durham, North Carolina
  - Oklahoma City, Oklahoma
  - Nashville, Tennessee
  - Houston, Texas
  - Burlington, Vermont
  - Chesapeake, Virginia
- Canada (4):
  - Kamloops, British Columbia
  - London, Ontario
  - Toronto, Ontario
  - Montreal, Quebec

REFERENCES:
- [Derived] Locatelli F, Spasovski G, Dimkovic N, Wanner C. Long-Term Evaluation of Colestilan in Chronic Kidney Disease Stage 5 Dialysis Patients with Hyperphosphataemia. Blood Purif. 2016;41(4):247-53. doi: 10.1159/000441648. Epub 2015 Dec 16. PMID 26670307

RESULTS

PARTICIPANT FLOW:
Groups:
- MCI-196: 3, 6, 9, 12, or 15 g/ day as titrated
Period: Overall Study
Arm/Group | MCI-196
Started | 116
Completed | 61
Not Completed | 55
Not completed — Adverse Event | 19
Not completed — Death | 6
Not completed — Lack of Efficacy | 4
Not completed — Physician Decision | 5
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 10
Not completed — Other Reasons | 10

BASELINE CHARACTERISTICS:
Arm/Group | MCI-196
Number analyzed (Participants) | 116
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (13.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40
  Male | 76

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Events (AE)
Time Frame: 52 weeks
Measure: Number; unit: participants
Arm/Group | MCI-196
Number analyzed (Participants) | 116
participants
  At least 1 treatment-emergent AE | 109
  At least 1 drug-related treatment-emergent AE | 50
  At least 1 treatment-emergent serious AE | 63

2. Secondary Outcome: The Change in Serum Phosphorus From Baseline to Week 52
Time Frame: 52 weeks
Population: Intent-to-treat (ITT) with last observation carried forward (LOCF). (ITT population included all enrolled subjects who took at least one dose of study medication and had at least one post-enrollment efficacy value after the start of study medication.)
Measure: Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | MCI-196
Number analyzed (Participants) | 116
mg/dL | -1.18 (2.05) [-1.56 to -0.81]

ADVERSE EVENTS:
Time Frame: 52 weeks
Arm/Group | MCI-196
Serious Adverse Events (participants affected / at risk) | 63/116
Other Adverse Events (participants affected / at risk) | 106/116
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCI-196 (N=116)
Hypertensive crisis (Vascular disorders) | 3
Arteriosclerosis obliterans (Vascular disorders) | 1
Haemorrhage (Vascular disorders) | 1
Jugular vein thrombosis (Vascular disorders) | 1
Malignant hypertension (Vascular disorders) | 2
Superior vena caval occlusion (Vascular disorders) | 1
Vena cava thrombosis (Vascular disorders) | 1
Accelerated hypertension (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Venous stenosis (Vascular disorders) | 1
Peripheral vascular disorder (Vascular disorders) | 1
Deep vein thrombosis (Vascular disorders) | 2
Hypotension (Vascular disorders) | 2
Steal syndrome (Vascular disorders) | 1
Pyrexia (General disorders) | 3
Catheter related complication (General disorders) | 3
Non-cardiac chest pain (General disorders) | 3
Chest pain (General disorders) | 1
Ascites (Gastrointestinal disorders) | 1
Pneumatosis intestinalis (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Diarrhoea (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Mallory-Weiss syndrome (Gastrointestinal disorders) | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1
Bacteraemia (Infections and infestations) | 2
Pharyngeal abscess (Infections and infestations) | 1
Diabetic foot infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 7
Sepsis (Infections and infestations) | 6
Gastroenteritis (Infections and infestations) | 2
Urinary tract infection (Infections and infestations) | 5
Wound infection staphylococcal (Infections and infestations) | 1
Wound infection (Infections and infestations) | 1
Escherichia urinary tract infection (Infections and infestations) | 1
Gangrene (Infections and infestations) | 3
Peritonitis bacterial (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 3
Bacterial sepsis (Infections and infestations) | 1
Arteriovenous graft site infection (Infections and infestations) | 1
Helicobacter gastritis (Infections and infestations) | 1
Cardiac failure congestive (Cardiac disorders) | 7
Angina pectoris (Cardiac disorders) | 3
Coronary artery disease (Cardiac disorders) | 9
Cardiac discomfort (Cardiac disorders) | 1
Acute myocardial infarction (Cardiac disorders) | 2
Atrial fibrillation (Cardiac disorders) | 5
Myocardial ischaemia (Cardiac disorders) | 1
Angina unstable (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Cardiac arrest (Cardiac disorders) | 3
Atrial flutter (Cardiac disorders) | 1
Supraventricular tachycardia (Cardiac disorders) | 1
Fluid overload (Metabolism and nutrition disorders) | 5
Diabetic ketoacidosis (Metabolism and nutrition disorders) | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 6
Calciphylaxis (Metabolism and nutrition disorders) | 2
Electrolyte imbalance (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Acute pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Lupus nephritis (Renal and urinary disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Renal failure acute (Renal and urinary disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Renal cyst ruptured (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Femur fracture (Injury, poisoning and procedural complications) | 1
Tibia fracture (Injury, poisoning and procedural complications) | 1
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 3
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 1
Hip fracture (Injury, poisoning and procedural complications) | 1
In-stent coronary artery restenosis (Injury, poisoning and procedural complications) | 1
Vena cava injury (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Ammonia increased (Investigations) | 1
International normalised ratio increased (Investigations) | 1
Mental status changes (Psychiatric disorders) | 1
Drug abuse (Psychiatric disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 3
Pancytopenia (Blood and lymphatic system disorders) | 1
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 2
Transient ischaemic attack (Nervous system disorders) | 1
Lacunar infarction (Nervous system disorders) | 1
Metabolic encephalopathy (Nervous system disorders) | 1
Partial seizures (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 3
Carotid artery stenosis (Nervous system disorders) | 2
Prostate cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Gastrointestinal arteriovenous malformation (Congenital, familial and genetic disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MCI-196 (N=116)
Abdominal discomfort (Gastrointestinal disorders) | 7
Abdominal distension (Gastrointestinal disorders) | 1
Ascites (Gastrointestinal disorders) | 5
Diarrhoea (Gastrointestinal disorders) | 23
Flatulence (Gastrointestinal disorders) | 2
Impaired gastric emptying (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 24
Nausea (Gastrointestinal disorders) | 26
Abdominal pain (Gastrointestinal disorders) | 5
Oesophagitis (Gastrointestinal disorders) | 1
Reflux gastritis (Gastrointestinal disorders) | 1
Abdominal pain upper (Gastrointestinal disorders) | 1
Abdominal pain lower (Gastrointestinal disorders) | 2
Hypoaesthesia oral (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 11
Dyspepsia (Gastrointestinal disorders) | 10
Stomatitis (Gastrointestinal disorders) | 1
Haematochezia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 2
Faecaloma (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 2
Colitis (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 2
Abdominal adhesions (Gastrointestinal disorders) | 1
Diverticulum intestinal (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Polyp colorectal (Gastrointestinal disorders) | 1
Glossodynia (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Rectal haemorrhage (Gastrointestinal disorders) | 2
Umbilical hernia, obstructive (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2
Melaena (Gastrointestinal disorders) | 1
Oesophageal stenosis (Gastrointestinal disorders) | 1
Contusion (Injury, poisoning and procedural complications) | 2
Fall (Injury, poisoning and procedural complications) | 3
Haemodialysis-induced symptom (Injury, poisoning and procedural complications) | 13
Procedural hypertension (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula site complication (Injury, poisoning and procedural complications) | 11
Mouth injury (Injury, poisoning and procedural complications) | 1
Procedural dizziness (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 2
Arteriovenous fistula occlusion (Injury, poisoning and procedural complications) | 1
Excoriation (Injury, poisoning and procedural complications) | 3
Joint sprain (Injury, poisoning and procedural complications) | 1
Wound (Injury, poisoning and procedural complications) | 1
Arteriovenous graft site haemorrhage (Injury, poisoning and procedural complications) | 1
Procedural pain (Injury, poisoning and procedural complications) | 3
Vascular graft complication (Injury, poisoning and procedural complications) | 1
Venous injury (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Arteriovenous fistula aneurysm (Injury, poisoning and procedural complications) | 2
Arteriovenous fistula site haemorrhage (Injury, poisoning and procedural complications) | 4
Ulna fracture (Injury, poisoning and procedural complications) | 1
Limb injury (Injury, poisoning and procedural complications) | 1
Arteriovenous graft thrombosis (Injury, poisoning and procedural complications) | 3
Arteriovenous fistula thrombosis (Injury, poisoning and procedural complications) | 2
Procedural hypotension (Injury, poisoning and procedural complications) | 2
Post procedural complication (Injury, poisoning and procedural complications) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 11
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 13
Orthopnoea (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 4
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 2
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 1
Rhonchi (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 3
Chylothorax (Respiratory, thoracic and mediastinal disorders) | 1
Productive cough (Respiratory, thoracic and mediastinal disorders) | 2
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 3
Pleural rub (Respiratory, thoracic and mediastinal disorders) | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 2
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypercapnia (Respiratory, thoracic and mediastinal disorders) | 1
Lung infiltration (Respiratory, thoracic and mediastinal disorders) | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1
Delirium (Psychiatric disorders) | 1
Confusional state (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 9
Stress (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 4
Drug abuse (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 2
Herpes zoster (Infections and infestations) | 1
Lower respiratory tract infection (Infections and infestations) | 1
Clostridial infection (Infections and infestations) | 3
Pulmonary tuberculosis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 8
Cellulitis (Infections and infestations) | 2
Gangrene (Infections and infestations) | 2
Localised infection (Infections and infestations) | 1
Nail infection (Infections and infestations) | 1
Osteomyelitis (Infections and infestations) | 1
Gastroenteritis (Infections and infestations) | 3
Bronchitis (Infections and infestations) | 6
Nasopharyngitis (Infections and infestations) | 11
Sinusitis (Infections and infestations) | 1
Enterococcal infection (Infections and infestations) | 2
Postoperative wound infection (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 9
Bacterial disease carrier (Infections and infestations) | 1
Subcutaneous abscess (Infections and infestations) | 1
Arteriovenous fistula site infection (Infections and infestations) | 3
Tooth abscess (Infections and infestations) | 1
Clostridium difficile colitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Furuncle (Infections and infestations) | 1
Peritonitis bacterial (Infections and infestations) | 1
Ear infection (Infections and infestations) | 1
Hepatitis C (Infections and infestations) | 1
Onychomycosis (Infections and infestations) | 1
Catheter related infection (Infections and infestations) | 1
Catheter site infection (Infections and infestations) | 1
Pleural infection bacterial (Infections and infestations) | 1
Staphylococcal infection (Infections and infestations) | 2
Graft infection (Infections and infestations) | 1
Wound infection staphylococcal (Infections and infestations) | 1
Oral candidiasis (Infections and infestations) | 1
Oesophageal candidiasis (Infections and infestations) | 1
Muscle tightness (Musculoskeletal and connective tissue disorders) | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 7
Neck pain (Musculoskeletal and connective tissue disorders) | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 8
Joint swelling (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 4
Muscle spasms (Musculoskeletal and connective tissue disorders) | 6
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Costochondritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 3
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Bursitis (Musculoskeletal and connective tissue disorders) | 1
Trigger finger (Musculoskeletal and connective tissue disorders) | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1
Groin pain (Musculoskeletal and connective tissue disorders) | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1
Post herpetic neuralgia (Nervous system disorders) | 1
Cerebrovascular accident (Nervous system disorders) | 1
Hemiparesis (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 3
Dizziness (Nervous system disorders) | 9
Headache (Nervous system disorders) | 11
Paraesthesia (Nervous system disorders) | 1
Facial palsy (Nervous system disorders) | 2
Syncope (Nervous system disorders) | 1
Dementia (Nervous system disorders) | 2
Somnolence (Nervous system disorders) | 1
Altered state of consciousness (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Aphasia (Nervous system disorders) | 1
Restless legs syndrome (Nervous system disorders) | 1
Carotid artery occlusion (Nervous system disorders) | 1
Carotid artery stenosis (Nervous system disorders) | 1
Pyrexia (General disorders) | 9
Chest discomfort (General disorders) | 3
Asthenia (General disorders) | 2
Malaise (General disorders) | 4
Oedema peripheral (General disorders) | 8
Chest pain (General disorders) | 4
Feeling hot (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Feeling cold (General disorders) | 1
Face oedema (General disorders) | 3
Fatigue (General disorders) | 2
Local swelling (General disorders) | 1
Localised oedema (General disorders) | 1
Chills (General disorders) | 4
Pain (General disorders) | 1
Influenza like illness (General disorders) | 2
Gait disturbance (General disorders) | 2
Catheter related complication (General disorders) | 1
Vessel puncture site haemorrhage (General disorders) | 1
Inflammation (General disorders) | 1
Catheter site pain (General disorders) | 1
Breath sounds abnormal (Investigations) | 3
Blood cholesterol increased (Investigations) | 1
Blood parathyroid hormone increased (Investigations) | 1
Methicillin-resistant staphylococcal aureus test positive (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Blood glucose increased (Investigations) | 1
Hepatic enzyme increased (Investigations) | 1
Blood phosphorus increased (Investigations) | 1
Venous pressure increased (Investigations) | 1
Ammonia increased (Investigations) | 1
Gram stain positive (Investigations) | 1
Weight decreased (Investigations) | 2
Vitamin D decreased (Investigations) | 1
Liver function test abnormal (Investigations) | 1
Cardiac murmur (Investigations) | 2
Blood creatine phosphokinase increased (Investigations) | 2
Chest X-ray abnormal (Investigations) | 1
Cardiovascular function test abnormal (Investigations) | 1
Activated partial thromboplastin time abnormal (Investigations) | 1
International normalised ratio abnormal (Investigations) | 1
Prothrombin time abnormal (Investigations) | 1
Electrocardiogram T wave abnormal (Investigations) | 1
Gamma-glutamyltransferase increased (Investigations) | 1
Prostatic specific antigen increased (Investigations) | 1
Blood glucose decreased (Investigations) | 2
Blood culture positive (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 14
Hypoglycaemia (Metabolism and nutrition disorders) | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 7
Hypocalcaemia (Metabolism and nutrition disorders) | 7
Hypokalaemia (Metabolism and nutrition disorders) | 4
Hyperhomocysteinaemia (Metabolism and nutrition disorders) | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Metabolic acidosis (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 2
Iron deficiency (Metabolism and nutrition disorders) | 1
Folate deficiency (Metabolism and nutrition disorders) | 2
Vitamin D deficiency (Metabolism and nutrition disorders) | 1
Hypernatraemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Hypervolaemia (Metabolism and nutrition disorders) | 2
Increased appetite (Metabolism and nutrition disorders) | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 5
Rash generalised (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5
Blister (Skin and subcutaneous tissue disorders) | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 1
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Periorbital oedema (Skin and subcutaneous tissue disorders) | 2
Post inflammatory pigmentation change (Skin and subcutaneous tissue disorders) | 1
Pruritus generalised (Skin and subcutaneous tissue disorders) | 2
Rash (Skin and subcutaneous tissue disorders) | 1
Rash pruritic (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 3
Urticaria (Skin and subcutaneous tissue disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Urinary tract disorder (Renal and urinary disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Polyuria (Renal and urinary disorders) | 1
Renal failure chronic (Renal and urinary disorders) | 1
Atrial fibrillation (Cardiac disorders) | 4
Bradycardia (Cardiac disorders) | 2
Angina pectoris (Cardiac disorders) | 5
Diastolic dysfunction (Cardiac disorders) | 1
Coronary artery occlusion (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 2
Atrioventricular block first degree (Cardiac disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Conduction disorder (Cardiac disorders) | 1
Bundle branch block left (Cardiac disorders) | 1
Cardiac tamponade (Cardiac disorders) | 1
Cardiomyopathy (Cardiac disorders) | 1
Atrial flutter (Cardiac disorders) | 1
Cardiomegaly (Cardiac disorders) | 2
Supraventricular tachycardia (Cardiac disorders) | 1
Mitral valve incompetence (Cardiac disorders) | 1
Tachyarrhythmia (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Hypotension (Vascular disorders) | 10
Hypertension (Vascular disorders) | 9
Orthostatic hypotension (Vascular disorders) | 2
Arteriosclerosis obliterans (Vascular disorders) | 1
Air embolism (Vascular disorders) | 1
Haematoma (Vascular disorders) | 1
Jugular vein distension (Vascular disorders) | 1
Vasodilatation (Vascular disorders) | 1
Venous occlusion (Vascular disorders) | 1
Peripheral arterial occlusive disease (Vascular disorders) | 1
Arterial thrombosis limb (Vascular disorders) | 1
Aortic dilatation (Vascular disorders) | 1
Scleral haemorrhage (Eye disorders) | 1
Eye swelling (Eye disorders) | 1
Ocular hyperaemia (Eye disorders) | 1
Conjunctivitis allergic (Eye disorders) | 1
Conjunctivitis (Eye disorders) | 1
Cataract (Eye disorders) | 1
Eye irritation (Eye disorders) | 1
Anaemia (Blood and lymphatic system disorders) | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Leukocytosis (Blood and lymphatic system disorders) | 1
Leukopenia (Blood and lymphatic system disorders) | 2
Atrial septal defect (Congenital, familial and genetic disorders) | 1
Hypothyroidism (Endocrine disorders) | 2
Hyperparathyroidism secondary (Endocrine disorders) | 2
Gallbladder polyp (Hepatobiliary disorders) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Seasonal allergy (Immune system disorders) | 2
Inner ear inflammation (Ear and labyrinth disorders) | 1
Sudden hearing loss (Ear and labyrinth disorders) | 1
Erectile dysfunction (Reproductive system and breast disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other